CLINICAL TRIAL: NCT03664921
Title: A Phase II Randomized, Double-Blind, Placebo-Controlled, Cross-Over Study Investigating the Safety and Efficacy of Omnitram in Diabetic Neuropathy
Brief Title: Omnitram Safety and Efficacy in the Treatment of Diabetic Neuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Syntrix Biosystems, Inc. (Industry)
Collaborators: DF/Net Research (Unknown); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Omni-Pain-201; 5R44DA040378-03 (NIH)
Record Dates: First submitted 2018-09-07; First posted 2018-09-11 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2020-09

CONDITIONS: Diabetic Neuropathies; Neuropathic Pain; Pain, Chronic
Keywords: Analgesia
MeSH Terms: conditions — Diabetic Neuropathies; Neuralgia; Chronic Pain; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Omnitram (Experimental): Oral Omnitram (10 mg tablets) dosed three times daily. During the first two weeks each dose will be titrated between 1 tablet (10 mg) and 4 tablets (40 mg) to provide pain relief. The doses administered at the end of two weeks will be maintained during the final two weeks of treatment.
  Interventions: Drug: Omnitram Oral Tablet
- Placebo (Placebo Comparator): Oral placebo (tablets) dosed three times daily. During the first two weeks each dose will be titrated between 1 tablet and 4 tablets to provide pain relief. The doses administered at the end of two weeks will be maintained during the final two weeks of treatment.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Omnitram Oral Tablet — Administered three times daily for 28 consecutive days.
  Arms: Omnitram
Drug: Placebo Oral Tablet — Administered three times daily for 28 consecutive days.
  Arms: Placebo

SUMMARY:
This study evaluates the analgesic effect of Omnitram for the treatment of painful diabetic neuropathy. Each subject with diabetic neuropathy will be treated for four weeks with Omnitram and for four weeks with placebo. The order of the Omnitram and placebo treatment will be random.

DETAILED DESCRIPTION:
A multi-centered, randomized, double-blind, placebo-controlled, two-period cross-over study to compare the safety and efficacy of Omnitram (30 mg to 120 mg daily) and placebo in patients with painful diabetic polyneuropathy. For subjects receiving treatment for neuropathic pain prior to study enrollment, their treatment will be tapered and stopped at least 2 weeks before they will be enrolled. Approximately fifty subjects will be randomized in a double-blind manner to a 4-week treatment period of Omnitram or placebo. After a washout of at least one week, patients will cross-over to the other treatment for a second 4 week treatment period with Omnitram or placebo.

During the first two weeks of each treatment period, guided by efficacy and tolerability, the dose will be increased from 3 tablets to 12 tablets per day given in three equal doses at approximately at 8 am, 2 pm and 8 pm (i.e., if the tablet is Omnitram, 30, 60, 90 or 120 mg/day). During the final two weeks of the treatment period, the doses will be kept constant at the highest tolerated titrated dose. Up to six tablets daily of 500 mg oral acetaminophen can be used as rescue medication except on the last 4 days of each treatment segment (Days 26, 27, 28, and 29).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between the ages of 18 and 75 years of age.
2. Diabetes mellitus diagnosis for at least 6 months.
3. Total glycosylated hemoglobin of <=12%.
4. Antidiabetic therapy used at screening will not be changed during the study.
5. Clinical diagnosis, confirmed by the Investigator, of painful diabetic neuropathy with symptoms and signs for at least 6 months.
6. Lower extremity pain, from diabetic neuropathy, present daily for the previous 3 months.
7. Patients currently requiring opioid treatment must be taking daily doses of an opioid-based analgesic equivalent to <=160mg of oral morphine.
8. Average neuropathic pain intensity over last 3 days before randomization (Segment 1, Study Day 1) of at least 4 on a 0-10 scale (0 = no pain; 10 = the worst possible pain).
9. Diabetic neuropathy confirmed by 1 of the following:

   * Clinical signs (distal sensory disturbance/lack of distal deep tendon reflexes).
   * Electrophysiological tests (slowing of nerve conduction or reduction of amplitude of sensory action potential).
   * Abnormal quantitative sensory testing (reduction or absence of pin sensibility and/or vibration sensibility on Total Neuropathy Score - Nurse (TNSn) examination in lower and/or upper extremities at screening.
10. Able and willing to give informed consent.
11. Able to comply with all study procedures.
12. If female, must not be of childbearing potential or must agree to use one or more of the following forms of contraception during screening and for 30 days following study drug dosing: hormonal (e.g., oral, transdermal, intravaginal, implant or injection); double barrier (i.e., condom, diaphragm with spermicide); intrauterine device (IUD) or system (IUS); vasectomized partner (6 months minimum); or abstinence; or bilateral tubal ligation (if no conception post-procedure).
13. Complete blood count (CBC) within normal range for the testing facility or not clinically significant.
14. Electrocardiogram (ECG), AST, ALT, and urinalysis values within the normal range for the testing facility or not clinically significant.
15. Normal renal function: Glomerular filtration rate (GFR) calculated by Cockcroft-Gault formula > 60 ml/min.
16. Negative pregnancy test within 1 week of Segment 1, Study Day 1.
17. Negative urine test for substances of abuse per CRU standards.
18. Negative serology tests for HIV, hepatitis B surface antigen, and hepatitis C virus antibody.
19. Body Mass Index (BMI) 19.0 to 40 kg/m.

Exclusion Criteria:

1. Clinically significant abnormal vital signs including oral temperature > 38°C or history of current illness.
2. Inability to exclude other causes of polyneuropathy including: alcoholism, vitamin B12 deficiency, endocrinopathies, vasculitides, heavy metal exposure, drug use, and malignancy (direct or paraneoplastic).
3. History of seizures, epilepsy, or recognized increase risk of seizure (e.g. head trauma, metabolic disorders, alcohol and drug withdrawal).
4. History of cirrhosis or laboratory evidence of liver disease.
5. Use of serotonergic drugs and drugs that impair serotonin metabolism (e.g., mirtazapine, trazodone); monoamine oxidase inhibitors, including linezolid, methylene blue; serotonin and norepinephrine reuptake inhibitors, except fluoxetine, within 14 days of Segment 1, Study Day 1 or during the study, use of fluoxetine within 28 days of Segment 1, Study Day 1, or during the study; and selective serotonin re-uptake inhibitors. Use of tricyclic antidepressants and other tricyclic drugs including cyclobenzaprine and promethazine; triptans; 5-HT3 receptor antagonists; neuroleptics. Use of benzodiazepines or other central nervous system depressants including non-benzodiazepine sedative hypnotics, anxiolytics, tranquilizers, muscle relaxants, general anesthetics, antipsychotics within 14 days of Segment 1, Study Day 1, or during the study. Use of opiates, including tramadol, within 28 days of Segment 1, Study Day 1, or during the study. Use of all other analgesics, except acetaminophen, within 14 days of Segment 1, Study Day 1, or during the study.
6. History of previous anaphylaxis, severe allergic reaction to tramadol, codeine or other opioid drugs.
7. Contraindication to use of opioids, tramadol, or acetaminophen.
8. Use of non-pharmacological pain therapy.
9. Any other unstable acute or chronic disease that could interfere with the evaluation of the safety of the study drug as determined by the principal Investigator in dialogue with the Sponsor's Medical Monitor.
10. Currently pregnant or breast-feeding a child.
11. Unlikely to comply with the study protocol.
12. Known or suspected alcohol or drug abuse within the past 12 months.
13. Received another investigational agent within 4 weeks before screening visit, or receiving any other investigational agent during this study.
14. Any concurrent disease or condition that in the opinion of the investigator impairs the subject's ability to complete the trial. Psychological, familial, sociological, geographical or medical conditions which, in the Investigator's opinion, could compromise compliance with the objectives and procedures of this protocol or obscure interpretation of the trial's data.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2020-08-17 (Actual); Study Completion 2020-08-17 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Scale | up to 28 days of each treatment.
  Subjects rate their pain intensity on a scale from 0 = no pain to 10 = worst possible pain

SECONDARY OUTCOMES:
Neuropathic Pain Symptom Inventory | The questionnaire is completed at Day 1 and Day 29 of both treatments.
  Subjects complete the questionnaire.
Sleep Problem Scale | The questionnaire is completed at Day 1 and Day 29 of both treatments.
  Subjects complete the questionnaire.
Major Depression Inventory | The questionnaire is completed at Day 1 and Day 29 of both treatments.
  Subjects complete the questionnaire.
Global Assessment of Treatment | The assessment is completed on Day 29 of both treatments.
  Independently the subject and Investigator assess the treatment on a 5-point scale (excellent, very good, good, fair, poor).
Global Impression of Change | The assessment is completed on Day 29 of both treatments.
  The subject assesses overall change on a 7-point scale (very much improved, much improved, minimally improved, no change, minimally worse, much worse, very much worse).
Average Daily Use of Acetaminophen | Day 1 through Day 25 of both treatments.
  Subjects may use a maximum of 3 grams of acetaminophen each day.
Adverse Events | Subjects report adverse events throughout study enrollment; investigators observe adverse events during subject clinic visits on Day 7 and Day 29 of each treatment, and at the final safety visit 2 weeks after the completing both treatments.
  Adverse events include: 1) reports by subjects; and 2) observations by investigators.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Kahn, MD, Study Director — Syntrix Biosystems
Locations (4):
- United States (4):
  - Orange County Research Institute, Anaheim, California
  - Core Healthcare Group, Cerritos, California
  - St. Louis Clinical Trials, St Louis, Missouri
  - Endeavor Clinical Trials, LLC, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No